CLINICAL TRIAL: NCT05511155
Title: Efficacy of Oxygen Therapy in Primary Headache Disorder
Brief Title: Oxygen Therapy for Headache
Status: Completed | Type: Observational
Sponsor: Aksaray University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ilker kacer, Medical Doctor, Aksaray University Training and Research Hospital
Other Study IDs: 64-SBKAEK
Record Dates: First submitted 2022-08-16; First posted 2022-08-22 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Primary Headache Disorder
Keywords: oxygen therapy; migraine; emergency department; cluster type headache
MeSH Terms: conditions — Headache Disorders, Primary; Migraine Disorders; Emergencies | interventions — Oxygen

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- O-15: 15 lt/min oxygen
  Interventions: Other: Oxygen therapy
- O-8: 8 lt/min oxygen
  Interventions: Other: Oxygen therapy
- A-15: 15 lt/min room air
  Interventions: Other: Oxygen therapy
- A-8: 8 lt/min room air
  Interventions: Other: Oxygen therapy

INTERVENTIONS:
Other: Oxygen therapy — Oxygen therapy will be given for 15 minutes with a non-rebreathing mask.

SUMMARY:
Headache is one of the common causes of emergency department admissions and constitutes approximately 2%. Although the exact mechanism is not clear, It is known that high-flow oxygen therapy is effective in headache treatment. There are limited studies related to the use of oxygen therapy in headaches and its derivatives in the literature. In this study, the investigators aimed to compare the high and medium flow oxygen therapies with placebo in primary headache disorders.

DETAILED DESCRIPTION:
Four different treatment methods were determined; 1) high-flow oxygen (15lt/min oxygen), 2) medium-flow oxygen (8lt/min oxygen), 3) high-flow room air as placebo (15 lt/min room air), 4) medium-flow room air as placebo (8 lt/min room air). All four treatment methods will be applied to all patients included in the study. One of the four treatments will be randomly applied at each separate ED admission with a gap of 1 week or more in between. This randomization will be performed by a computer at the time of admission. A study nurse will administer the patient's therapy according to the computer's current decision for 15 minutes. Patients and treating physicians will be blinded to the selected therapy. After 15 minutes of the end of treatment (at the 30th minute of the start of treatment), the treating physician will ask patients if they need rescue analgesia and analgesia will be administered if necessary. Additional analgesia is at the discretion of the treating physician. Patient data, including demographics, medical history, and findings of a physical examination performed before and after therapy will be recorded by the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* age 18-55 years
* frequent attacks of primary headache disorders according to International Headache Society (IHS) criteria

Exclusion Criteria:

* secondary headache disorders
* oxygen-dependent chronic illnesses such as chronic obstructive pulmonary disease
* a history of cerebrovascular disease
* pregnancy
* active smokers or living with a smoker.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: all patients had one to six headache attacks per month which were started before 50 years old and were present for more than one year.
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
visual analog scale score | 0-60 minutes
  primary endpoint is the relative reduction in visual analog scale (a psychometric response scale) score in the placebo versus oxygen group to determine whether there was a difference between the high-flow and mid-flow therapies. visual analog scale scaled from 0-100 points with 0 meaning "no pain" and 100 points meaning "worst possible pain".

SECONDARY OUTCOMES:
rescue analgesia | 30 th minutes
  rescue analgesia (yes/no)
length of stay | 0-300 minutes
  length of stay in the emergency department (time in minutes)
duration of a pain | 0-300 minutes
  duration of a pain attack (time in minutes)
readmission | 0-7 days
  readmission to the emergency department within 7 days (yes/no)

CONTACTS AND LOCATIONS:
Locations (1):
- Aksaray University Aksaray Training and Research Hospital, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedman BW, Grosberg BM. Diagnosis and management of the primary headache disorders in the emergency department setting. Emerg Med Clin North Am. 2009 Feb;27(1):71-87, viii. doi: 10.1016/j.emc.2008.09.005. PMID 19218020
- [Background] Roberto G, Raschi E, Piccinni C, Conti V, Vignatelli L, D'Alessandro R, De Ponti F, Poluzzi E. Adverse cardiovascular events associated with triptans and ergotamines for treatment of migraine: systematic review of observational studies. Cephalalgia. 2015 Feb;35(2):118-31. doi: 10.1177/0333102414550416. Epub 2014 Sep 22. PMID 25246519
- [Background] Mo H, Chung SJ, Rozen TD, Cho SJ. Oxygen Therapy in Cluster Headache, Migraine, and Other Headache Disorders. J Clin Neurol. 2022 May;18(3):271-279. doi: 10.3988/jcn.2022.18.3.271. PMID 35589316
- [Background] Petersen AS, Barloese MC, Lund NL, Jensen RH. Oxygen therapy for cluster headache. A mask comparison trial. A single-blinded, placebo-controlled, crossover study. Cephalalgia. 2017 Mar;37(3):214-224. doi: 10.1177/0333102416637817. Epub 2016 Jul 11. PMID 27013239